CLINICAL TRIAL: NCT06998368
Title: A Causal Role for Voltage-gated Cav1.2 Calcium Channels in Mediating 5G FR1 Effects on Sleep-associated Brain Health in Humans
Acronym: 5G Cav12 Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hans-Peter Landolt (Other)
Collaborators: Federal Office for the Environment, Switzerland (Other Government)
Responsible Party: Sponsor-Investigator, Hans-Peter Landolt, Prof. Dr. sc. nat., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 5G-Cav1.2 Sleep
Record Dates: First submitted 2025-04-23; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Mediation of 5G Effects on Sleep
Keywords: 5G; CACNA1C; CaV1.2; electromagnetic; EMF; nimodipine; RF-EMF; sleep; rs7304986; voltage-gated calcium channel; brain
MeSH Terms: interventions — Nimodipine

STUDY DESIGN:
Intervention Model Description: Each participant of the sleep study will undergo 4 experimental night recordings. On each of the experimental nights, one unique combination of two different interventions will be applied: active exposure to 5G RF-EMF or sham and administration of nimodipine (i.e. verum) or placebo.
  The four combinations will be:
  * placebo + sham exposure
  * placebo + active exposure
  * verum + sham exposure
  * verum + active exposure. The sequence order of the 4 nights conditions will be randomized.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (24):
- Arm2 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm1 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining eighteen sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm3 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm4 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm6 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm7 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm8 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm9 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm10 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm11 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm12 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm5 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm13 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm14 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm15 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm16 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm17 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm18 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm19 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm20 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm21 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm22 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm23 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF
- Arm24 (Other): The study includes 24 arms, each corresponding to one of the 24 unique sequences in which the four intervention combinations (drug/placebo × active/sham) can be administered. Given that the expected total sample size is 30 participants, six of these sequences will be randomly assigned to two participants, while the remaining 18 sequences will be assigned to one participant each.
  Interventions: Drug: Nimodipine Capsules; Radiation: 5G RF-EMF

INTERVENTIONS:
Drug: Nimodipine Capsules — Two times 30 mg nimodipine or placebo will be administered orally 45 minutes prior to the start of the 5G FR1 exposure. The verum and placebo capsules will look the same, in order to preserve the double-blinding.
Radiation: 5G RF-EMF — Participants will be exposed to a standardized electromagnetic field of the latest mobile radio standard (5G) or a sham field for 30 minutes on each of the experimental nights. The active field is characterized by 3.6 GHz frequency [TDD] with 100 MHz bandwidth, 12-14 Hz modulation and is comparable to a phone call with a commercially available, modern cell phone. Both the 5G and sham exposures are performed with the same exposure apparatus, according to a double-blind study design.

SUMMARY:
Electromagnetic fields (EMFs) generated by the use of 5G technology influence certain sleep characteristics, especially in individuals carrying a specific genetic variant of a protein in the brain that regulates the activity of nerve cells. This protein is a voltage-gated calcium channel called CaV1.2 and could be involved in the effects of 5G technology on sleep. The calcium channel CaV1.2 can be selectively blocked by the drug nimodipine.

To demonstrate that CaV1.2 is indeed involved in the effects of 5G technology on sleep, the researchers are investigating in this study, with healthy subjects carrying the sought-after genetic variant, whether the administration of nimodipine and thus the blockade of the calcium channel before exposure mitigates or eliminates the effects of EMF on sleep health.

DETAILED DESCRIPTION:
This study tests a causal role of voltage-gated CaV1.2 calcium channels in mediating the effects of a 5G electromagnetic field on sleep-related brain health in humans.

The study comprises a large-scale genetic screening in order to select the allele-carriers, a sleep screening night, and four experimental nights where participants are exposed to either an active 5G field or sham, combined with either nimodipine (which is a brain-penetrant L-type calcium channel blocker) or placebo. Participants will undergo polysomnographic recordings, high-density electroencephalography (EEG) during wake, peripheral measurements, cognitive and neuropsychiatric assessments.

ELIGIBILITY:
Inclusion Criteria:

For the first part of the study (genotyping and questionnaires):

* Age: 20-40 years old.
* German and/or English language skills (reading and writing)
* Informed Consent as documented by signature

For the second and third party of the study:

* Completion of the first part of the present study or of the precursor study (BASEC-ID: 2016-02049)
* CACNA1C rs7304986 T/C allele-carrier
* Male gender
* Female gender if using hormonal contraception for the duration of the study (e.g., pill as combination/single preparation, three-month injection, hormonal IUD, hormonal implant, hormonal patch)
* Right-handedness
* Body Mass Index (BMI): BMI comprised between 17.0 kg/m2 and 26.0 kg/m2

  * Moderate alcohol consumption (less than 5 reported alcoholic drinks per week)
  * Moderate caffeine consumption (less than 3 reported caffeinated beverage or food products per day such as cola, coffee, energy drinks, green and black tea, chocolate)
  * Informed Consent as documented by signature.

Exclusion Criteria:

For the second and third party of the study:

* Travel with a time difference of more than 2 time zones in the last 30 days before study entry or during the study period
* Shift work at night
* Extreme chronotype or duration of sleep (5 hours < reported habitual sleep duration per night > 10 hours)
* Known sleep disorders or diseases
* Serious acute or chronic neurological, mental, or general medical conditions that, in the opinion of the investigator, may pose a risk to participation or affect study measurements
* Use of medications (regularly or during the study period) that, in the opinion of the investigator, may affect study measurements.
* Use of illegal drugs
* Smoking (or other tobacco use)
* Known or suspected non-compliance with the investigators' indications
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc.
* Severe skin allergies or hypersensitivities
* Participation in another clinical trial in the last 30 days prior to inclusion or during the present study
* Contraindications to nimodipine, e.g., known hypersensitivity or allergy to nimodipine or any of the excipients
* Other cases in which the use of nimodipine is discouraged according to the summary of product characteristics (SPC)
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Lack of safe contraception, defined as: female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases (Note: Female participants who are surgically sterilized / hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential)
* Sleep apnea and nocturnal myoclonus index of ≥ 5 per hour of sleep (as assessed during the screening night)
* Sleep efficiency < 80% (as assessed during the screening night)
* Other relevant findings in the screening/adaptation night (e.g., indications of sleep disorders), which in the opinion of the investigator may pose a risk for participation or influence the study measurements.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sleep spindle center frequency | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions
  In previous research, the investigators detected a positive shift in the sleep spindle center frequency (during NREM sleep phase) after 30-min pre-sleep exposure to a 5G signal at 3600 MHz, 100 MHz bandwidth in heterozygous T/C allele-carriers (rs7304986) compared to sham.
  The sleep spindle center frequency is a parameter that can be extracted from the overnight electroencephalographic recordings.

SECONDARY OUTCOMES:
Sex distribution of participants | At the large-scale genetic screening
  Self-reported biological sex (male or female) is recorded during the large-scale genetic screening (first study part) via an online questionnaire.
Age of Participants | At the large-scale genetic screening
  Age is recorded in years based on the year of birth provided during the large-scale genetic screening (first study part) via an online questionnaire.
Pregnancy status | At the large-scale genetic screening
  Female participants report current pregnancy status during the large-scale genetic screening (first study part) via an online questionnaire.
EEG power spectra during Non-Rapid-Eye-Movement (NREM) sleep | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions
  Power spectra will be computed from artifact-free EEG data recorded during NREM sleep. Spectral power (µV²/Hz) will be computed in standard frequency bands.
Total sleep time | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions
  Sleep electroencephalographic data allow to extract total sleep time (min) (total amount of time spent asleep)
Neurocognitive performance as assessed in the psychomotor vigilance task (PVT) | Assessed on each of the four experimental nights, pre- and post-sleep
  The PVT is administered before and after sleep at each experimental night and provides a score reflecting sustained or vigilant attention performance.
Heart rate | Assessed on each of the four experimental nights, from electrocardiographic recordings during pre-sleep exposure and polysomnographic overnight recordings
  Heart rate (bpm) is extracted from electrocardiographic recording during exposure and from polysomnographic overnight recordings
Handedness of participants | At the large-scale genetic screening
  Participants report their handedness (right-handed or left-handed) during the large-scale genetic screening (first study part) via an online questionnaire.
BMI of participants | At the large-scale genetic screening
  Self-reported height (in centimeters) and weight (in kilograms) of participants is reported during the large-scale genetic screening (first study part) via an online questionnaire. From Height and Weight, BMI is calculated.
Highest level of education of participants | At the large-scale genetic screening
  The highest level of education of participants (elementary school, professional school, high school, university of applied sciences and arts, or university) is self-reported during the large-scale genetic screening (first study part) via an online questionnaire.
Phone call time | At the large-scale genetic screening
  Participants report their phone call time without headphones (Not at all, Less than 1 hour per week, 1-2 hours per week or more than 2 hours per week) during the large-scale genetic screening (first study part) via an online questionnaire.
Caffeine consumption | At the large-scale genetic screening
  Participants report their caffeine consumption (None, 1-2 caffeinated foods or beverages per day, 3-5 caffeinated foods or beverages per day or More than 5 caffeinated foods or beverages per day) during the large-scale genetic screening (first study part) via an online questionnaire.
Alcohol consumption | At the large-scale genetic screening
  Participants report their alcohol consumption (None, Less than 1 glass per week, 1-2 glasses per week, 3-5 glasses per week or More than 5 glasses per week) during the large-scale genetic screening (first study part) via an online questionnaire.
Electrohypersensitivity (EHS) status | At the large-scale genetic screening
  Participants report their EHS status during the large-scale genetic screening (first study part) via filling out the online questionnaire by M. Röösli, E. Mohler, and P. Frei (2010).
Sleep disturbances | At the large-scale genetic screening
  The presence of sleep disturbances is self-reported by participants during the large-scale genetic screening (first study part) via an online questionnaire.
Comorbidities | At the large-scale genetic screening
  Participants self-report the presence of comorbidities during the large-scale genetic screening (first study part) via an online questionnaire.
Night-shift work | At the large-scale genetic screening
  Participants report if they engage in night shift work during the large-scale genetic screening (first study part) via an online questionnaire.
Use of medications | At the large-scale genetic screening
  Self-reported use of medication is recorded during the large-scale genetic screening (first study part) via an online questionnaire.
Use of illegal drugs | At the large-scale genetic screening
  Self-reported use of illegal drugs is recorded during the large-scale genetic screening (first study part) via an online questionnaire.
Use of tobacco products | At the large-scale genetic screening
  Use of tobacco products is reported during the large-scale genetic screening (first study part) via an online questionnaire.
Subjective sleep quality | At the large-scale genetic screening
  Participants report about their subjective sleep quality during the large-scale genetic screening (first study part) via filling out the online questionnaire "Pittsburgh Sleep Quality Index" (high global PSQI score indicates poor sleep quality).
Daytime sleepiness | At the large-scale genetic screening
  Participants report about their daytime sleepiness during the large-scale genetic screening (first study part) via filling out the online questionnaire "Epworth Sleepiness Scale " (high ESS score indicates high daytime sleepiness).
Diurnal preference | At the large-scale genetic screening
  Participants report about their diurnal preference during the large-scale genetic screening (first study part) via filling out the online questionnaire "Munich Chronotype Questionnaire" (if the mid-sleep time on the MCTQ is earlier than 04:00, the participant is considered as preferential morning type, otherwise as preferential evening type).
Habitual bedtime | At the large-scale genetic screening
  Participants report about their subjective habitual bedtime (hh:mm) during the large-scale genetic screening (first study part) via filling out the online questionnaire "Pittsburgh Sleep Quality Index".
Habitual rise time | At the large-scale genetic screening
  Participants report about their subjective habitual rise time (hh:mm) during the large-scale genetic screening (first study part) via filling out the online questionnaire "Pittsburgh Sleep Quality Index".
Reported time to fall asleep | At the large-scale genetic screening
  Participants report about their subjective time to fall asleep (min) during the large-scale genetic screening (first study part) via filling out the online questionnaire "Pittsburgh Sleep Quality Index".
Reported sleep duration | At the large-scale genetic screening
  Participants report about their subjective sleep duration (h:mm) during the large-scale genetic screening (first study part) via filling out the online questionnaire "Pittsburgh Sleep Quality Index".
Positive and Negative Affect Schedule | At the large-scale genetic screening
  Participants report about positive and negative feelings (over the last 12 months) during the large-scale genetic screening (first study part) via filling out the online questionnaire "Positive and Negative Affect Schedule".
Nocturnal mentation | At the large-scale genetic screening
  Participants report about their nocturnal mentation during the large-scale genetic screening (first study part) via filling out online the "Dream Thought Questionnaire".
Depressive tendency | At the large-scale genetic screening
  Participants report about their depressive-like symptoms (experienced in the last 2 weeks) during the large-scale genetic screening (first study part) via filling out the online questionnaire "Beck Depression Index II (BDI-II)".
Mental suggestibility tendency | At the large-scale genetic screening
  Participants report about their mental suggestibility tendency during the large-scale genetic screening (first study part) via filling out the online questionnaire "Short Suggestibility Scale".
Schizotypal tendency | At the large-scale genetic screening
  Participants report about their schizotypal tendencies during the large-scale genetic screening (first study part) via filling out an online adaptation of the questionnaire "Magical Ideation Scale (MIS)".
ADHD tendency | At the large-scale genetic screening
  Participants report about their ADHD-like symptoms during the large-scale genetic screening (first study part) via filling out the online questionnaire "Adult ADHD Self-Report Scale v1.1 (ASRS)".
EEG power spectra during wakefulness | Assessed on each of the four experimental nights, from pre- and post-sleep wake electroencephalographic recordings
  Power spectra will be computed from artifact-free EEG data recorded during wakefulness. Spectral power (µV²/Hz) will be computed in standard frequency bands.
EEG power spectra during Rapid Eye Movement (REM) sleep | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions
  Power spectra will be computed from artifact-free EEG data recorded during REM sleep. Spectral power (µV²/Hz) will be computed in standard frequency bands.
Aperiodic component of the EEG power spectrum during NREM sleep | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions
  The NREM sleep power spectra will be used to extract and parametrize the aperiodic component.
Aperiodic component of the EEG power spectrum during REM sleep | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions
  The REM sleep power spectra will be used to extract and parametrize the aperiodic component.
Aperiodic component of the EEG power spectrum during wakefulness | Assessed on each of the four experimental nights, from pre- and post-sleep wake electroencephalographic recordings
  The wake power spectra will be used to extract and parametrize the aperiodic component.
Periodic component of the EEG power spectrum during NREM sleep | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions
  Gaussian peaks detected in the NREM sleep power spectrum will be used to extract the periodic components, including center frequency, power, and bandwidth.
Periodic component of the EEG power spectrum during REM sleep | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions.
  Gaussian peaks detected in the REM sleep power spectrum will be used to extract the periodic components, including center frequency, power, and bandwidth.
Periodic component of the EEG power spectrum during wakefulness | Assessed on each of the four experimental nights, from pre- and post-sleep wake electroencephalographic recordings
  Gaussian peaks detected in the wake power spectrum will be used to extract the periodic components, including center frequency, power, and bandwidth.
Sleep efficiency | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions
  Sleep electroencephalographic data allow to extract sleep efficiency (%) ((total sleep time/time in bed) * 100)
Sleep latency | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions.
  Sleep electroencephalographic data allow to extract sleep latency (time between lights-off and first occurrence of NREM sleep stage N2).
Wakefulness after sleep onset | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions
  Sleep electroencephalographic data allow to extract WASO (min) (wakefulness after sleep onset).
Time spent in the different sleep stages | Assessed on each of the four experimental nights, from overnight electroencephalographic recordings following randomized combinations of drug (nimodipine or placebo) and RF-EMF exposure (5G or sham), with a minimum of 3 days washout between sessions
  Sleep electroencelographic data allow to calculate the time (min) spent in each sleep substage (NREM1, NREM2, NREM3, REM).
Neurocognitive performance as assessed in the sequential finger tapping task (FTT) | Assessed on each of the four experimental nights, pre- and post-sleep
  The FTT is administered before and after sleep at each experimental night and provides a score reflecting procedural memory and learning performance.
Neurocognitive performance as assessed in the visuospatial 2D Object Location Task (OLT) | Assessed on each of the four experimental nights, pre- and post-sleep
  The OLT is administered before and after sleep at each experimental night and provides a score reflecting declarative memory and learning performance.
Heart rate variability | Assessed on each of the four experimental nights, from electrocardiographic recordings during pre-sleep exposure and polysomnographic overnight recordings
  Heart rate variability is extracted from electrocardiographic recording during exposure and from polysomnographic overnight recordings.
Pupil size | Assessed on each of the four experimental nights, from pupillometry recordings during pre-sleep exposure.
  Pupil size variation is recorded during exposure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Institute of Pharmacology and Toxicology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Any disclosure of information to individuals not directly involved in the study must be approved by the owner of the data.

REFERENCES:
- See also: Pre-print of our previous research project, providing the background for the current study — https://www.medrxiv.org/content/10.1101/2024.12.16.24319082v1